CLINICAL TRIAL: NCT06110975
Title: Deprescribing dRugs for Overactive Bladder in the Elderly in General Practice - a Randomized Controlled Trial With a Nested Mixed Methods Study
Brief Title: Deprescribing dRrugs for Overactive Bladder in General Practice (DROP)
Acronym: DROP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Estrup Olesen (Other)
Collaborators: University College of Northern Denmark (Other)
Responsible Party: Sponsor-Investigator, Anne Estrup Olesen, Professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: K2023-012
Record Dates: First submitted 2023-10-05; First posted 2023-11-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Overactive Bladder; Deprescribing; PIMS
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Primary care clinics are randomized to the deprescribing intervention or control group. The control group is not contacted and comparison relies on register data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The primary care clinics in the intervention group will contact and evaluate all patients receiving one or more of the following drugs:
  G04BD04 Oxybutynin G04BD07 Tolterodine G04BD08 Solifenacin G04BD09 Trospium G04BD10 Darifenacine G04BD11 Fesoterodine G04BD12 Mirabegron The patients will be asked to discontinue the treatment and eventually be deprescribed
  Interventions: Other: deprescribing-intervention
- Control group (No Intervention): The primary care clinics in the control group will not contact and evaluate patients and are not informed about the study. Data will be extracted from registries

INTERVENTIONS:
Other: deprescribing-intervention — The clinical guideline on "Deprescribing drugs for OAB" in The North Denmark Region serves as the basis for the intervention. The guideline provides recommended procedures for the deprescribing process. The guideline offers procedures for the deprescribing process and includes a deprescribing algorithm and a symptom questionnaire designed to evaluate the impact of medications utilized in the treatment of OAB.
  Other Names: DROB (Deprescribing dRugs for Overactive Bladder)
  Arms: Intervention group

SUMMARY:
The objective is to understand and evaluate the effectiveness of a deprescribing intervention in primary care, specifically targeting medications for overactive bladder in individuals aged 65 or older.

DETAILED DESCRIPTION:
Potentially inappropriate medication is prescribed medications with an unfavorable risk-benefit profile, for which there might be better, safer, or more cost-effective alternatives. Anticholinergic drugs for Overactive Bladder (OAB) is an example of a potentially inappropriate medication in the elderly, calling for attention and possible deprescribing. Due to their crucial role in maintaining a patient's medication regimen, primary care settings are widely regarded as the optimal location for conducting medication reviews and deprescribing interventions.

This study utilizes a mixed methods explanatory sequential design, nested in a randomised controlled trial to explore deprescribing drugs for Overactive Bladder (OAB). General practices will be randomized into two groups. The intervention group will then be evaluated in a mixed methods setup and finish the study with a comparison to the control group. The mixed methods approach employs a quantitative approach following the intervention group and investigates the prevalence of deprescribing the drugs in question. Secondly, a qualitative approach will be used to delve into the experiences of general practitioners (GPs), support staff, and patients during the deprescribing process. Finally, the quantitative and qualitative findings are merged to gain a comprehensive understanding of deprescribing for OAB. This integrated approach enhances insights and informs future interventions and recommendations. After the mixed methods studies are completed the control group will be used in an overall comparison of the two groups using registry data

ELIGIBILITY:
Inclusion Criteria:

* patient must have been prescribed one of the following drugs for OAB within the last 14 months
* patient must be able to speak and understand Danish

Exclusion Criteria:

* too cognitively impaired to participate or otherwise unfit to participate as estimated by general practitioner
* receiving neurological or urogenital ambulatory care for their overactive bladder symptoms

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Difference in proportion of patients receiving drugs for overactive bladder | 6 months
  The primary outcome will be the difference in the proportion of patients receiving drugs for overactive bladder before and after a 6-month follow-up period.

SECONDARY OUTCOMES:
proportion of patients in the intervention group who had deprescribing initiated but not sustained | 6 months
  Descriptive characteristics of the proportion of patients in the intervention group who had deprescribing initiated but not sustained.
The proportion of patients where deprescribing was not initiated | 6 months
  Descriptive characteristics of the proportion of patients in the intervention group where deprescribing was not initiated.
Changes and distribution of bladder symptoms | 6 months
  Descriptive characteristics and distribution of bladder symptoms between and within the groups before and after the intervention

OTHER OUTCOMES:
A qualitative score measuring experiences | Approximately 6 months after the study initiates
  Interviews to explore how GPs, staff members, and patients have experienced the intervention and which strategies have been used for the successful deprescribing of drugs for overactive bladder to understand when and how the algorithm is useful using thematic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Olesen, Professor, Principal Investigator — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Soerensen AL, Haase Juhl M, Krogh ML, Gronkjaer M, Kristensen JK, Olesen AE. Deprescribing as a Way to Reduce Inappropriate Use of Drugs for Overactive Bladder in Primary Care (DROP): Protocol for a Cluster Randomized Controlled Trial With an Embedded Explanatory Sequential Mixed Methods Study. JMIR Res Protoc. 2024 Jul 23;13:e56277. doi: 10.2196/56277. PMID 39042875